CLINICAL TRIAL: NCT01426308
Title: Method Comparison and Clinical Specificity Study: Evaluation of the Infinium HD Cytogenetic Abnormality Test
Status: Completed | Type: Observational
Sponsor: Illumina, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Cyto-001
Record Dates: First submitted 2011-08-29; First posted 2011-08-31 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2011-09

CONDITIONS: Post-natal Cytogenetics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Method Comparison Group: The method comparison group will consist of de-identified, leftover DNA samples from patients referred for post-natal cytogenetic testing.
- Clinical Specificity Group: The clinical specificity group will consist of de-identified, leftover DNA samples from non-phenotypic patients, or patients not referred for post-natal cytogenetic testing.

SUMMARY:
The study will determine the performance of the Infinium HD Test.

* The primary objective of the study is to assess the performance of the Infinium HD Test using banked DNA samples extracted from whole blood patient samples derived from the intended use population.
* The secondary objective of the study is to determine the background number of chromosomal abnormalities per person in the general population based on the resolution of the Infinium HD Test.

ELIGIBILITY:
Method Comparison - Sample Inclusion Criteria

The following are criteria for inclusion of extracted genomic DNA samples in the method comparison sample pool:

1. Sample is from a patient referred for post-natal cytogenetic testing.
2. Sample gender is known.
3. Sample quantity available for testing is ≥ 1 microgram of genomic DNA at a concentration of 60-80 nanograms per microliter (60-80ng/µl).
4. Sample is extracted genomic DNA from EDTA or heparin-anticoagulated whole blood.
5. Sample has been stored at 2 to 8°C or -15 to -25°C for no greater than three years from the date of extraction.
6. Sample has been tested by a reference method. Acceptable reference methods include karyotype, FISH, qPCR, MLPA, and methylation analysis.

Method Comparison - Sample Exclusion Criteria

1. Sample is from a patient not referred for post-natal cytogenetic testing.
2. Sample is from a patient referred for cytogenetic oncology testing.
3. Sample quantity < 1 microgram of genomic DNA or less than 60 nanograms per microliter (60ng/µl).
4. Sample was improperly stored or was extracted from a sample that was improperly stored.
5. Sample was tested by an Illumina array during standard of care testing.

Clinical Specificity - Sample Inclusion Criteria

The following are criteria for inclusion of extracted genomic DNA samples in the clinical specificity sample pool:

1. Sample gender is known.
2. Sample is from a patient not referred for post-natal cytogenetic testing.
3. Sample quantity available for testing is ≥ 1 microgram of genomic DNA at a concentration of at least 60-80 nanograms per microliter (60-80ng/µl).
4. Sample is extracted genomic DNA from EDTA or heparin-anticoagulated whole blood.
5. Sample has been stored at 2 to 8°C or -15 to -25°C for no greater than three years from the date of extraction.

Clinical Specificity - Sample Exclusion Criteria

1. Sample is from a patient referred for post-natal cytogenetic testing.
2. Sample quantity < 1 microgram of genomic DNA or less than 60 nanograms per microliter (60ng/µl).
3. Sample was improperly stored or was extracted from a sample that was improperly stored.

Min Age: 1 Minute | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Leftover, de-identified DNA extracted from EDTA or heparin anticoagulated whole blood samples.
Sampling Method: Probability Sample
Enrollment: 900 (Actual)
Dates: Start 2011-08; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor College of Medicine, Houston, Texas
  - ARUP Laboratories, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No